CLINICAL TRIAL: NCT01989442
Title: Efficacy and Safety of Nasal Mask and Prong Use in Non-invasive Ventilation for Newborns
Brief Title: Nasal Mask and Prong Use in Non-invasive Ventilation for Newborns
Acronym: NIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Ufuk Cakir, MD, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Map-NIV Trial
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: cpap failure; bronchopulmonary dysplasia; nasal trauma; ventilation duration; non-invasive ventilation
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal Mask (Experimental): patients who receive NIV by nasal mask interface after randomization
  Interventions: Device: nasal mask
- nasal prong (Active Comparator): patients who receive NIV by nasal prongs as interface after randomization
  Interventions: Device: binasal prongs

INTERVENTIONS:
Device: binasal prongs — patients randomized to binasal prongs for NIV will use binasal prongs as an interface during continuous positive airway pressure support
  Other Names: viasys healthcare infant flow system- binasal prongs
  Arms: nasal prong
Device: nasal mask — patients randomized to nasal mask for NIV will use nasal mask as an interface during continuous positive airway pressure support
  Other Names: viasys healthcare infant flow system-nasal mask
  Arms: Nasal Mask

SUMMARY:
The study aims to investigate efficacy and safety of nasal mask and prongs used in non-invasive ventilation in newborns by using esophageal pressure transducer.

The parameters including ventilation duration, hospitalization duration, pulmonary outcomes and side effects will be evaluated.

DETAILED DESCRIPTION:
Although it seems as more non-invasive there is still lack of data especially on efficacy of nasal mask use in NIV for newborns. By using esophageal pressure transducers we will evaluate the pressure supplied by the ventilation mode and compare it with more commonly used nasal prongs. The investigators will test the hypothesis of equivalence of nasal mask in comparison to prongs with better safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* all newborns who require NIV as first line treatment as respiratory support in delivery room or neonatal intensive care unit

Exclusion Criteria:

* who are intubated in delivery room or neonatal intensive care unit before randomization
* with congenital anomaly
* patients who require NIV more than 3 days

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
failure of NIV | 1 year
  patients who require endotracheal intubation after NIV treatment

SECONDARY OUTCOMES:
ventilation duration | 3 days
  both NIV and mechanical ventilation durations will be evaluated

OTHER OUTCOMES:
bronchopulmonary dysplasia | 1 year
  oxygen or pressure requirement on postmenstrual 36 weeks of gestational age
septal trauma rate | 1 year
  any destruction on nose that require treatment after use of NIV

CONTACTS AND LOCATIONS:
Overall Officials: Saadet ARSAN, Professor, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] McCarthy LK, Twomey AR, Molloy EJ, Murphy JF, O'Donnell CP. A randomized trial of nasal prong or face mask for respiratory support for preterm newborns. Pediatrics. 2013 Aug;132(2):e389-95. doi: 10.1542/peds.2013-0446. Epub 2013 Jul 29. PMID 23897911
- [Background] Kieran EA, Twomey AR, Molloy EJ, Murphy JF, O'Donnell CP. Randomized trial of prongs or mask for nasal continuous positive airway pressure in preterm infants. Pediatrics. 2012 Nov;130(5):e1170-6. doi: 10.1542/peds.2011-3548. Epub 2012 Oct 22. PMID 23090339